CLINICAL TRIAL: NCT03620123
Title: A Randomized Phase II Study on the OPTimization of IMmunotherapy in Squamous Carcinoma of the Head and Neck
Acronym: OPTIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-KHT-0117; 2017-003349-14 (EudraCT Number); CA209-998 (Other: Bristol-Myers Squibb GmbH & Co. KGaA)
Record Dates: First submitted 2018-07-13; First posted 2018-08-08 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck; Carcinoma, Squamous Cell of Head and Neck
Keywords: SCCHN; Nivolumab; Ipilimumab
MeSH Terms: conditions — Recurrence; Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Ipilimumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab and Ipilimumab (Experimental): Nivolumab 3 mg/kg of body weight intravenous infusion every two weeks and ipilimumab 1 mg/kg of body weight intravenous infusion every six weeks
  Interventions: Drug: Nivolumab and Ipilimumab
- Docetaxel (Other): docetaxel 75 mg/m² intravenous infusion every three weeks
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Nivolumab and Ipilimumab — Nivolumab 3 mg/kg of body weight intravenous infusion every two weeks and ipilimumab 1 mg/kg of body weight intravenous infusion every six weeks
  Arms: Nivolumab and Ipilimumab
Drug: Docetaxel — docetaxel 75 mg/m² intravenous infusion every three weeks
  Arms: Docetaxel

SUMMARY:
AIO-KHT-0117 (OPTIM) is a phase II, open-label randomized, multicenter study of nivolumab and ipilimumab on the optimization of immunotherapy in squamous carcinoma of the head and neck after prior platinum-based therapy.

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter, phase II trial. Patients with recurrent or metastatic squamous cell carcinoma of the head and neck will be enrolled in this trial will initiate palliative systemic treatment with nivolumab monotherapy (240 mg fixed dose Q2W). Tumor response will be assessed after 4, 8, 12, 18 and 24 weeks to capture early progressors. Patients with (radiologic) tumor progression during the first 6 months of NIVO mono will be randomized (1:1) to receive either docetaxel (75 mg/m2 Q3W) or nivolumab+ipilimumab combination (Nivolumab 3mg/kg Q2W + Ipilimumab 1mg/kg Q6W) until progressive disease [PD] or death. Patients without PD within 6 months NIVO monotherapy continue treatment under study surveillance for a maximum of 12 months measured from first dose of NIVO or until documented disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent including participation in translational research and any locally required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥ 18 years at time of study entry
3. Histological or cytological confirmed recurrent or metastatic squamous cell carcinoma of the head and neck (HNSCC) or nasal sinus not amenable to local therapies
4. Availability of tumor tissue from biopsy for determination of PD-L1 and HPV status according to the following priority ranking: i) recent biopsy (≤3 months old) without intervening therapy; ii) any recent biopsy (≤3 months old); iii) any archival tumor tissue (> 3 months old) [Biopsy should be excisional, incisional or core biopsy. Fine needle aspiration is not allowed.]
5. Progression or recurrence during or after platinum-based palliative chemotherapy for relapsed or metastatic disease OR Progression within 6 months after completion of definitive platinum-containing radiochemotherapy for locally advanced disease
6. At least 1 measurable lesion according to RECIST 1.1
7. ECOG performance status 0-1
8. Completion of local therapy for brain metastases with discontinuation of steroids prior to start of study treatment
9. Adequate blood count, liver enzymes, and renal function

   * neutrophil count > 1.5 x 10^6/mL
   * platelet count ≥ 100 x 10^9/L (>100,000 per mm³)
   * hemoglobin ≥ 9 g/dL
   * INR ≤ 1.5 and PTT ≤ 1.5 x lower limit during the last 7 days before therapy
   * AST (SGOT)/ALT (SGPT) < 3 x institutional upper limit of normal (5 x lower limit in case of liver metastases)
   * bilirubin < 1.5 x ULN
   * serum creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 40 mL/min
10. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
11. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. [WOCBP should use an adequate method to avoid pregnancy for 5 months (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of nivolumab.] Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) do not require contraception.
12. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. [Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of up to 7 months after the last dose of IMP.] Men who are not of childbearing potential (ie, surgically sterile or azoospermic ) do not require contraception
13. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Nasopharynx carcinoma or carcinoma of salivary glands
2. Life expectancy less than 3 months
3. Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results, including but not limited to:

   1. Minor surgery ≤ 24 hours prior first dose of nivolumab monotherapy
   2. Anticancer treatment during the last 30 days prior to start of nivolumab monotherapy, including systemic therapy, or major surgery [palliative radiotherapy has to be completed at least 2 weeks prior to start of nivolumab monotherapy]
   3. Known active HBV, HCV or HIV infection
   4. Active tuberculosis
   5. Any other active infection requiring systemic therapy
   6. History of allogeneic tissue/solid organ transplant (including hematopoietic stem cell transplantation)
   7. Diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of nivolumab-monotherapy or randomization.
   8. Has an active autoimmune disease requiring systemic treatment within the past 3 months before enrolment or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study. Psoriasis not requiring treatment is not excluded from the study.
   9. Live vaccine within 30 days prior to the first dose of nivolumab-monotherapy or during study treatment.
   10. Other active malignancy requiring treatment
   11. Clinically significant or symptomatic cardiovascular/cerebrovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) within 6 months before enrollment
   12. History or clinical evidence of CNS metastases

   Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria:
   * are asymptomatic and
   * have no requirement for steroids 6 weeks prior to start of nivolumab-monotherapy. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS metastases
4. Medication that is known to interfere with any of the agents applied in the trial.
5. Has known hypersensitivity to nivolumab or ipilimumab or docetaxel or any of the constituents of the products.
6. Any other efficacious cancer treatment except protocol specified treatment at study start.
7. Patient has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. [Subjects with ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study.]
8. Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner].
9. Prior therapy with an anti-Programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-Programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand,a member of the Tumor Necrosis Factor Receptor [TNFR] family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
10. Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer
11. Previous treatment in the present study (does not include screening failure) [Criterion is not applicable during re-assessment of eligibility for randomization].
12. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
13. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2022-06-19 (Actual)

PRIMARY OUTCOMES:
objective response rate in all randomized subjects | approx. 48 months

SECONDARY OUTCOMES:
overall survival [OS] | approx. 48 months
Progression-free survival [PFS] | approx. 42 months
Best overall response [BOR] | approx. 42 months
Duration of Response [DOR] | approx. 42 months
Health related quality of life | approx. 42 months
  EORTC QLQ-C30
Health related quality of life: EORTC QLQ-H&N35 | approx. 42 months
  EORTC QLQ-H&N35
Health related quality of life: EQ-5D-5L | approx. 42 months
  EQ-5D-5L
Toxicity/Safety according to CTC-AE-criteria | approx. 42 months

OTHER OUTCOMES:
Tumor tissue analysis | approx. 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Grünwald, Prof. Dr., Principal Investigator — Essen University Hospital
Locations (1):
- Essen University Hospital, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de
- See also: AIO-Studien-gGmbH — http://www.aio-studien-ggmbh.de